CLINICAL TRIAL: NCT06329323
Title: SerUm and Plasma MicroRNAs in Malignant Ovarian gERm Cell Tumours
Acronym: SUMMER
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 23CX8477
Record Dates: First submitted 2023-12-04; First posted 2024-03-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Germ Cell Ovarian Cancer; Germ Cell Tumor; Germ Cell Cancer; Germ Cell Neoplasia; Ovary Cancer; Ovary Neoplasm; Ovarian Cancer; Ovarian Neoplasms
Keywords: Germ Cell Cancer; microRNA; miRNA; Ovarian Cancer
MeSH Terms: conditions — Ovarian Germ Cell Cancer; Neoplasms, Germ Cell and Embryonal; Ovarian Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma (microRNA expression); tumour specimen (microRNA expression)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cases- Malignant Ovarian Germ Cell Tumour - Arm 1: Patients with a diagnosis of stage 1a MOGCT. Bloods taken at the following time points: Day 0, then 4 weeks; 6 months; 12 months; 24 months post-operatively
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Pathology specimen miRNA expression
- Cases - Malignant Ovarian Germ Cell Tumour - Arm 2: Patients with a diagnosis of stage 1b/1c MOGCT. Bloods taken at the following time points: Day 0, then 4 weeks; 6 months; 12 months; 24 months post-operatively OR post-final dose of adjuvant chemotherapy
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Pathology specimen miRNA expression
- Cases - Malignant Ovarian Germ Cell Tumour - Arm 3: Patients with a diagnosis of stage 2 or higher MOGCT. Bloods taken at the following time points: Day 0, then 4 weeks post-neoadjuvant chemotherapy, then 4 weeks; 6 months; 12 months; 24 months post-operatively
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Pathology specimen miRNA expression
- Controls - Benign Ovarian Germ Cell Tumour: Bloods taken at the time of diagnosis of BOGCT (single blood test)
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Pathology specimen miRNA expression
- Controls - No Known Gynaecological Pathology: Single blood test
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Serum and plasma microRNA quantification
Diagnostic Test: Pathology specimen miRNA expression — Pathology specimen mirNA expression - ALL MOGCT; OPTIONAL for BOGCT
  Groups: Cases - Malignant Ovarian Germ Cell Tumour - Arm 2; Cases - Malignant Ovarian Germ Cell Tumour - Arm 3; Cases- Malignant Ovarian Germ Cell Tumour - Arm 1; Controls - Benign Ovarian Germ Cell Tumour

SUMMARY:
The goal of this observational case-control study is to learn about the circulating and tissue microRNA expression, imaging and radiomic profiles of malignant ovarian germ cell tumours (MOGCT) compared to patients with a benign OGCT and no ovarian pathology.

The main question[s] it aims to answer are:

1. To understand the circulating miRNA expression of malignant ovarian germ cell tumours (MOGCTs) compared to those with benign ovarian germ cell tumours (BOGCTs)
2. To understand the imaging profile of MOGCTs compared to that of BOGCTs
3. To establish the relationship between serum and plasma miRNA expression in response to treatment and relapse of disease
4. To discover if miRNA expression correlates with radiomic features of OGCTs on both ultrasound and MRI
5. To see if we can link the micro RNAs in tumour samples to those found in blood samples, and to find a plausible explanation for why these micro RNAs are raised (in terms of the tumour biology itself).aims

Participants will have serial blood tests at different time points in their care to assess how circulating miRNA levels are affected by treatment and/or remission and/or relapse. If they have surgery, a pathology sample will be taken from the main tumour specimen. Radiomic analysis will take place on existing ultrasound images of their mass.

Researchers will compare the circulating miRNA profile of patients with a benign ovarian germ cell tumour and no ovarian pathology to see where the differences lie. If a patient with a BOGCT requires surgery, a pathology sample will be taken from the main tumour specimen. Radiomic analysis will take place on existing ultrasound images of their benign mass.

DETAILED DESCRIPTION:
Case population (MOGCTs):

1. Serum aFP (alpha fetoprotein), hCG (human chorionic gonadotrophin), LDH (lactate dehydrogenase) and Ca125 (cancer antigen 125) tumour markers measured at time of diagnosis
2. Additional serum and plasma sample to be obtained at the same time as initial bloods
3. Subsequent serum and plasma samples to be obtained as per study arms 1-3 based on cancer staging
4. Tissue samples will be obtained at the time of surgery

Control population:

Participants acting as controls will be identified from those attending for TV-USS where either a benign teratoma or no pathology is identified (e.g. from a gynaecology clinic). A total of 26ml of blood will be taken. Serum aFP, hCG, LDH and Ca125 will be measured as per routine clinical practice in patients with a benign OGCT.

Patients in the control population (benign germ cell tumours or patients with no known gynaecological pathology) will have a single blood test for miRNA analysis.

If participants require an operation for the benign GCT, tissue samples will be obtained at the time of surgery.

miRNA analysis will be performed using NanoString for the discovery panel. Further targeted sequencing will be performed in the larger prospective study using specific miRNA panels. This may be done using NanoString or a custom MiRNA assay primer.

Endpoint The pilot will be completed after the final patient has completed 12 months of follow up. The pilot data analysis will take place at that point.

We anticipate that the study will end 12 months after the final participant has completed 24 months of follow up, which gives 12 months for analysis of the samples. The number of participants to take part will be based on a power calculation performed at the time of analysis of the pilot data.

DATA COLLECTION AND MANAGEMENT Patients will enter study arm 1-3 based on cancer staging, or will belong to the control group.

Each participant will be followed up for a maximum of 2 years after they receive their definitive treatment (surgery and/or (neo)adjuvant chemotherapy). We anticipate this will be a maximum of 30 months total time in the study.

An interim analysis of data will be performed at 12 months, with a view to:

1. Identify key miRNAs for prospective validation
2. Allow for appropriate power calculation of the prospective validation study

ELIGIBILITY:
Inclusion Criteria:

* All patients with a new diagnosis of a malignant ovarian germ cell tumour.
* The control population will include all patients with a new diagnosis of a benign ovarian germ cell tumour or no known gynaecological pathology.

Exclusion Criteria:

* Previous or ongoing chemotherapy for MOGCT
* Previous surgery for MOGCT
* Pregnancy - this will be verbally communicated for those not having surgery or chemotherapy, for those having surgery or chemotherapy a urine pregnancy test should be negative and documented in the clinical notes.
* Fetal circulating DNA is known to be present in maternal blood and therefore pregnant women should not be included in this study
* Denial of informed consent
* Age <16 years
* History of any other cancer

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women aged over 16 with a diagnosis of a malignant ovarian germ cell tumour, benign ovarian germ cell tumour or no known gynaecological pathology may take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-04-14 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Difference in microRNA expression (plasma) between benign and malignant masses | 24 months
  Comparison of heatmaps based on mean expression of clusters across samples
Difference in microRNA expression (serum) between benign and malignant masses | 24 months
  Comparison of heatmaps based on mean expression of clusters across samples
microRNA expression (plasma) | 24 months
  Differential expression of microRNAs (assessed using a moderated t statistic and P values adjusted for multiple testing)
microRNA expression (serum) | 24 months
  Differential expression of microRNAs (assessed using a moderated t statistic and P values adjusted for multiple testing)

SECONDARY OUTCOMES:
Quantitative measure of circulating miRNA before treatment | 24 months
  miRNA expression in plasma samples of women with a diagnosis of a MOGCT compared to those of women with BOGCTs using nCounter miRNA Expression panels
Quantitative measure of circulating miRNA before treatment | 24 months
  miRNA expression in serum samples of women with a diagnosis of a MOGCT compared to those of women with BOGCTs using nCounter miRNA Expression panels
Quantitative measure of circulating miRNA after treatment | 24 months
  miRNA expression in plasma samples of women with a diagnosis of a MOGCT compared to those of women with BOGCTs using nCounter miRNA Expression panels
Quantitative measure of circulating miRNA after treatment | 24 months
  miRNA expression in serum samples of women with a diagnosis of a MOGCT compared to those of women with BOGCTs using nCounter miRNA Expression panels
Performance of segmentation model on ultrasound images | 24 months
  Correlation between identification of region of interest (ROI) to examiner segmentation. Dice surface coefficient (DICE).
Performance of segmentation model on MRI images | 24 months
  Correlation between identification of region of interest (ROI) to examiner segmentation. Dice surface coefficient (DICE)
Performance of classification model on ultrasound images | 24 months
  Correlation between benign or malignant diagnosis by model vs ultrasound subjective assessment or histopathological diagnosis (area under the ROC curve (AUC), F1-score)
Performance of classification model on MRI images | 24 months
  Correlation between benign or malignant diagnosis by model vs ultrasound subjective assessment or histopathological diagnosis (area under the ROC curve (AUC), F1-score)

CONTACTS AND LOCATIONS:
Overall Officials: Srdjan Saso, PhD MRCOG MRCS, Principal Investigator — Imperial College Healthcare NHS Trust

IPD SHARING:
Plan to Share IPD: No